CLINICAL TRIAL: NCT06969612
Title: A Prospective, Phase IB Clinical Study on the Efficacy and Safety of Golidocitinib Combined With Tislelizumab and Chemotherapy as First-line Treatment for Advanced NSCLC
Brief Title: A Study on the Efficacy and Safety of Golidocitinib Combined With Tislelizumab and Chemotherapy as First-line Treatment for Advanced NSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Zhuo MingLei, Peking University Cancer Hospital & Institute, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025YJZ14
Record Dates: First submitted 2025-04-26; First posted 2025-05-14 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Pemetrexed; Cisplatin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Golidocitinib combined with tislelizumab and chemotherapy (Experimental): Take tislelizumab and chemotherapy for 2 cycles; and then take tislelizumab for 2 cycles and golidocitinib for 6 weeks; after cycle 5, patients receive tislelizumab and chemotherapy until the patients were intolerant or the disease progressed.
  Interventions: Drug: Tislelizumab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Albumin Paclitaxel; Drug: Golidocitinib

INTERVENTIONS:
Drug: Tislelizumab — 200 mg, intravenously on Day 1, every 3 weeks
Drug: Pemetrexed — administered via IV infusion
Drug: Cisplatin — administered via IV infusion
Drug: Carboplatin — administered via IV infusion
Drug: Paclitaxel — administered via IV infusion
Drug: Albumin Paclitaxel — administered via IV infusion
Drug: Golidocitinib — 75mg, once a day orally

SUMMARY:
The goal of this clinical trial is to learn if golidocitinib combined with tislelizumab and chemotherapy works in advanced NSCLC with PD-L1≥1%. The main question it aims to answer is:

Does the combination of golidocitinib with tislelizumab and chemotherapy can prolong the progression-free survival of patients with advanced NSCLC?

Participants will： Take tislelizumab and chemotherapy for 2 cycles; and then take tislelizumab and golidocitinib for 2 cycles; after cycle 5, patients receive tislelizumab and chemotherapy until the patients were intolerant or the disease progressed.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide the informed consent form with signatures and signing dates, including compliance with the requirements and restrictions listed in the informed consent Form (ICF) and this protocol;
2. At the time of signing the ICF, the age must be at least 18 years old, with no gender restrictions.
3. The ECOG score is 0 or 1.
4. Life expectancy ≥ 3 months;
5. Histological or cytological examination confirms that the newly diagnosed NSCLC is locally advanced (IIIB/C) or metastatic (stage IV) that cannot undergo radical surgery or radiotherapy;
6. PD-L1(22C3) ≥1%;
7. At least one measurable lesion (RECIST v1.1);
8. The bone marrow reserve and organ system functional reserve are sufficient, which can be summarized as follows:

   - Under the condition of not receiving growth factor support, the absolute neutrophil count (ANC) was ≥ 1.5×109/L.

   - Under the condition of not receiving growth factor support or blood transfusion, platelet count ≥ 100×109/L.

   - In the absence of blood transfusion or reception of erythropoietin, hemoglobin ≥ 9 g/dL.

   -Total bilirubin ≤ 1.5 × ULN; If one has Gilbert syndrome (unconjured hyperbilirubinemia), the total bilirubin should be ≤ 3 × ULN.

   -ALT and AST≤ 2.5 × ULN. For patients with recorded liver metastases, the levels of AST and ALT are ≤ 5 × ULN.

   -Blood creatinine ≤ 1.5 × ULN, or creatinine clearance rate calculated by the Cockcroft-Gault method ≥ 50 mL/min, or urine creatinine clearance rate measured within 24 hours ≥ 50 mL/min.
9. For patients with central nervous system metastases, the following conditions must be met before they can be enrolled:

   - No neurological symptoms or stable symptoms for at least 2 weeks after local treatment, no need to use corticosteroids or antiepileptic drugs, and hormone therapy should be discontinued within 3 days before the administration of the first study drug;
   * If the brain metastases have received local treatment (radiotherapy or surgery), there should be a time window of ≥2 weeks before the first administration of the study treatment to ensure that the adverse events related to local treatment have been reduced to CTCAE ≤ grade 1.
10. Women of Childbearing Potential (WOCBP) must undergo a urine and/or serum (if the urine test cannot be confirmed as negative) pregnancy test within 7 days before the first medication, and the result must be negative; WOCBP or the male and his WOCBP partner should agree to take effective contraceptive measures from the date of signing the ICF until 6 months after using the last dose of the study drug.

Exclusion Criteria:

1. Histology of lung adenocarcinoma confirmed the presence of EGFR19 deletion or L858R mutation and ALK, ROS-1 fusion gene mutation (non-adenocarcinoma patients are not required to undergo mandatory genetic testing).
2. Have received systemic chemotherapy, biological therapy, targeted therapy or immunotherapy for metastatic or advanced NSCLC before;
3. Interstitial pneumonia/immune pneumonia or interstitial changes are known to exist;
4. Subjects with known meningeal metastases, brainstem metastases, spinal cord metastases and/or compression, or active CNS metastases;
5. Have any of the following medical histories:

   * Currently participating in intervention clinical research and treatment, any drug still in the research and development stage needs to be eluted for 5 half-lives (or discussed with the research team);
   * Palliative radiotherapy has been received within 2 weeks before the first administration. Radiotherapy for more than 30% of the bone marrow or extensive radiotherapy needs to be completed within 4 weeks before administration.
   * Currently receiving (or unable to discontinue use at least one week before the first administration) drugs, herbal supplements, and foods that are known to be potent inducers or potent inhibitors of CYP3A Before the first administration, there were adverse events of CTCAE > grade 1 caused by the previous treatment (except for any degree of alopecia);
6. Have received solid organ or blood system transplants (such as having received allogeneic bone marrow transplants in the past or having received whole blood transfusions within 120 days of sample collection during the study period);
7. Subjects with severe pulmonary function decline (i.e., any FEV1 or DLCO < 60% of the predicted value). Previous interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid hormone therapy, current interstitial lung disease with active clinical symptoms (including interstitial changes in the lungs), immune pneumonia of grade 3 or above caused by immunotherapy, or treatment termination;
8. There is an active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, corticosteroids or immunosuppressants) within 2 years prior to the first administration. Alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency, etc.) are not regarded as systemic treatment;
9. Diagnosed with immune deficiency or undergoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days prior to the first administration of the study, the use of physiological doses of glucocorticoids (≤10 mg/ day prednisone or equivalent drugs) is permitted;
10. Diagnosed with other malignant tumors within 5 years prior to the first administration, excluding cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma and/or carcinoma in situ that has been evaluated as clinically cured;
11. Live vaccines, including attenuated live vaccines, have been administered within 30 days before the first administration (day 1 of Cycle 1), except for inactivated vaccines.
12. The researchers judged it as active tuberculosis, such as a positive tuberculin (PPD) test (induration diameter > 10 mm), a positive T-SPOT test, tuberculosis foci found on chest X-ray plain film /CT, or other positive results found based on clinical routine screening (except for those who have recovered after standardized anti-tuberculosis treatment as evaluated by the researchers);
13. Subjects with active infections, including but not limited to hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV); 1) Active HCV and HIV infection, that is, the corresponding antibody test result is positive; 2) Untreated active hepatitis B, defined as HBsAg positive with HBV DNA ≥1000IU/ml, or HBcAb positive with HBV DNA ≥1000IU/ml; However, research participants who meet the following conditions can also be enrolled: Before the first administration, if HBsAg was positive and HBV DNA was < 1000IU/ml, the study participants should receive anti-HBV treatment throughout the study treatment period to prevent viral reactivation.

13. For those with negative HBsAg, positive HBcAb and HBV DNA < 1000IU/ml, the participants of the study should have HBV DNA tested throughout the treatment period of the study.

14. Allergy to the drugs used in the research or their components; 15. Dysphagia, or suffering from active digestive system diseases, or having undergone major digestive tract surgeries, which may significantly affect the administration or absorption of the investigational drug (such as ulcerative lesions, inability to swallow drugs, uncontrollable nausea, vomiting, diarrhea and malabsorption syndrome); 16. Those that the researcher deems unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to ~24 months
  PFS is defined as the time from the first dose until the first documentation of progression or death from any cause, whichever occurs first, as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to ~24 months
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR), as assessed by the investigator using RECIST v1.1.
Disease Control Rate (DCR) | Up to ~24 months
  DCR is defined as the percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD), as assessed by the investigator using RECIST v1.1.
Duration of Response (DOR) | Up to ~24 months
  DOR is defined as the time from the first occurrence of a objective response to the time of documented disease progression, or death from any cause, whichever comes first, as assessed by the investigator using RECIST v1.1
Time To Response (TTR) | Up to ~24 months
  TTR is defined as the time from the first dose to the first time of documented objective response, as assessed by the investigator using RECIST v1.1 in participants with documented objective responses
Overall Survival (OS) | Up to ~60 months
  OS is defined as the time from first dose until the date of death due to any cause
Adverse events | Through study completion, an average of 2 year
  Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) and immune-related adverse events (irAEs), which includes laboratory tests, physical exams, electrocardiogram results and vital signs, according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No